CLINICAL TRIAL: NCT05598684
Title: Assessment of Predictive Factors for Persistence of Treatment After Initiation of Adalimumab With a Biosimilar (Adalimumab Fresenius KaBI or Substitution of Reference Adalimumab With the Fresenius Kabi Adalimumab Biosimilar in Patients With Chronic Inflammatory Diseases
Brief Title: SAPHIR : Assessment of Predictive Factors for Persistence of Treatment After Initiation of Adalimumab With a Biosimilar (Adalimumab Fresenius KaBI or Substitution of Reference Adalimumab With the Fresenius Kabi Adalimumab Biosimilar in Patients With Chronic Inflammatory Diseases
Acronym: SAPHIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fresenius Kabi, France (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A00946-37
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2023-07

CONDITIONS: Crohn Disease; Ulcerative Colitis; Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: Adult patients who agreed to initiate treatment with a biosimilar (adalimumab FK) or to replace the reference adalimumab with the adalimumab FK biosimilar

SUMMARY:
A prospective, longitudinal, multicentre, observational cohort follow-up study conducted in France.

DETAILED DESCRIPTION:
In a population of adult patients who are targeted to initiate adalimumab or previously treated with Humira® to get switched to a biosimilar (FK adalimumab) and followed up for a period of 12 months under routine medical practice conditions.

* Primary objective: to define predictive factors for the persistence of treatment
* Secondary objectives:

  * To assess the therapeutic benefit and the tolerability of the treatment
  * To describe the reasons for treatment discontinuations occurring during follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or over
* Patient who have been informed of the objectives and the conditions of the study and who did not object to its participation
* Patient diagnosed with one chronic inflammatory rheumatological (rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis) or chronic inflammatory bowel (Crohn's disease, ulcerative colitis) diseases
* Patient for whom the investigator has decided, with patient's agreement and prior to inclusion:
* Or to initiate adalimumab by prescribing a biosimilar (Adalimumab FK)
* Either to replace Humira® with a biosimilar (AdalimumabFK)

Exclusion Criteria:

* Patient enrolled in an interventional therapeutic trial at the time of inclusion
* Patient refusing or unable to comply with the study follow-up procedures (patient not contactable by telephone, unable to complete the self-administered questionnaire, or having poor French language skills, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with adalimumab for chronic inflammatory rheumatism (CIR) or inflammatory bowel disease (IBD).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Persistence of the biosimilar | Month 12
  Persistence of the biosimilar is defined as the maintenance of FK adalimumab for the twelve-month study period
Discontinuation of the biosimilar | Month 12
  Discontinuation of the biosimilar is defined as the definitive cessation of FK adalimumab

SECONDARY OUTCOMES:
Clinical status | Day 0
  Clinical Global Impression (CGI)-severity scale graded from 0 to 7 (0 is not evaluated, 1 is the best case and 7 the worst case)
Maintenance of therapeutic benefit | Month 6
  Clinical Global Impression (CGI)-improvement scale graded from 0 to 7 (0 is not evaluated, 1 is the best case and 7 the worst case)
Maintenance of therapeutic benefit | Month 12
  Clinical Global Impression (CGI)-improvement scale graded from 0 to 7 (0 is not evaluated, 1 is the best case and 7 the worst case)
Treatment acceptance | Day 0
  Acceptance of the chronic treatment assessed on D0 using the Accept® questionnaire
Quality of life assessment | Month 12
  Medical Outcome Study Short Form 12 (MOS SF-12) or "Short Form 12 " (SF-12) scale
Emotional state | Month 12
  Screening for symptoms of anxiety and depression involves the use of the HAD questionnaire.
Tolerability evaluation | Month 12
  Collection of all adverse events (serious or non serious)

CONTACTS AND LOCATIONS:
Locations (91):
- France (89):
  - Nouvelle Clinique BONNEFON, Alès
  - Ch Amiens Nord, Amiens
  - Chu Amiens Picardie Site Sud, Amiens
  - Cabinet Médical, Argeles
  - Ch Armentieres, Armentières
  - CH d'ARDECHE MERDIONALE, Aubenas
  - Cabinet de Gastroentérologie, Bayonne
  - Cabinet Médical, Besançon
  - Chu Besancon Hopital Jean Minjoz, Besançon
  - Clinique du Cèdre, Bois-Guillaume
  - AP HP Ambroise PARE, Boulogne-Billancourt
  - Ch Boulogne Sur Mer, Boulogne-sur-Mer
  - Hôpital Privé SAINT-MARTIN, Caen
  - Centre Consultations Polyclinique St Jean, Cagnes-sur-Mer
  - Ch Cahors, Cahors
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Clinique du Parc, Castelnau-le-Lez
  - Ch Chateauroux, Châteauroux
  - Cabinet Médical, Chilly-Mazarin
  - CHU CLERMONT FERRAND, site ESTAING, Clermont-Ferrand
  - Chu Gabriell Monpied, Clermont-Ferrand
  - AP HP Hôpital BEAUJON, Clichy
  - Ch Sud Francilien, Corbeil-Essonnes
  - Clinique Claude BERNARD, Ermont
  - Chu Grenoble Sud, Échirolles
  - Ch Annecy Genevois, Épagny
  - Centre Gastro Loire, Gien
  - Ch Haguenau, Haguenau
  - Cabinet Médical, La Madeleine
  - Forum Médica, Lattes
  - Ch Chartres Louis Pasteur, Le Coudray
  - Cabinet Médical Groupe, Le Folgoët
  - AP HP Hôpital BICETRE, Le Kremlin-Bicêtre
  - Cabinet Médical de Rhumatologie, Lézignan-Corbières
  - Chu Dupuytren 2, Limoges
  - Ch Bretagne Sud, Lorient
  - Medipole de La Meurthe - Cabinet Médical, Lunéville
  - Cabinet Médical TILSITT, Lyon
  - Hopital Prive Jean Mermoz Cabinet Medica, Lyon
  - Maison Médicale, Marolles-en-Brie
  - Centre Mutualiste LA FEUILLERAIE, Marseille
  - AP HM Hôpital NORD, Marseille
  - Cabinet de Rhumatologie, Mennecy
  - Ch Montauban, Montauban
  - Clinique PONT DE CHAUME, Montauban
  - MIMOUNE, Montereau-Fault-Yonne
  - Ghi Le Raincy Montfermeil, Montfermeil
  - Chu Hôtel Dieu, Nantes
  - Institut Des Mici-Clinique Ambroise Paré, Neuilly-sur-Seine
  - Cabinet Médical, Nice
  - Chu Nice Hôpital Pasteur, Nice
  - AP HP Hôpital LARRIBOISIERE, Paris
  - AP HP Hôpital SAINT ANTOINE, Paris
  - Cabinet Médical, Paris
  - Ap Hp Gh Pitie Salpetriere, Paris
  - Chu Cochin, Paris
  - Chu Bichat, Paris
  - Ch Lyon Sud, Pierre-Bénite
  - Cabinet Médical, Poissy
  - Cabinet Médical, Poitiers
  - Clinique CROIX du SUD, Quint-Fonsegrives
  - Hôpital Robert DEBRE, Reims
  - Chu Pontchaillou, Rennes
  - Cabinet Médical, Rodez
  - Cabinet Médical, Saint-Amand-les-Eaux
  - Hôpital St-Avold Groupe Sos Santé, Saint-Avold
  - Chu Saint Etienne Hôpital Nord, Saint-Etienne
  - Cabinet Médical, Saint-Louis
  - Hôpital d'Instruction des Armées BEGIN, Saint-Mandé
  - Cabinet Médical, Sarreguemines
  - Cabinet Médical, Strasbourg
  - Ch Strasbourg Hôpital Hautepierre, Strasbourg
  - Nouvel Hôpital Civil, Strasbourg
  - Ch Tarbes Lourdes, Tarbes
  - Hôpital Bel Air, Thionville
  - Cabinet Médical, Toulon
  - HIA Hôpital SAINT-ANNE, Toulon
  - CHU PURPAN Hôpital PIERRE PAUL RIQUET, Toulouse
  - Chu Rangueil, Toulouse
  - Clinique PASTEUR, Toulouse
  - Clinique MEDIPOLE GARONNE, Toulouse
  - Cabinet Médical, Tourcoing
  - Centre Rééd. Fonct. Trestel - Ch Lannion, Trévou-Tréguignec
  - Hpda Site Clinique Générale, Valence
  - Cabinet de Rhumatologie, Valenciennes
  - Cabinet Médical, Vannes
  - Ghm Les Portes Du Sud, Vénissieux
  - Ch Villeneuve Pôle de Sante Villeneuvois, Villeneuve-sur-Lot
  - Cabinet Médical, Villeurbanne
- Cabinet Médical, Pointe-à-Pitre, Guadeloupe
- Cabinet Médical, Saint-Pierre, Martinique